CLINICAL TRIAL: NCT03749876
Title: A Randomized Cross-over Clinical Trial of Unfiltered Cigarettes
Brief Title: A Study of Unfiltered Cigarettes Among Committed Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: California State University, San Marcos (Other); Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Eyal Oren, Associate Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TRDRP Award #580582
Record Dates: First submitted 2018-11-17; First posted 2018-11-21 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Cigarette Smoking; Tobacco Smoking
Keywords: Cigarette filters; Cigarette smoking; Unfiltered cigarettes
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research staff performing the statistical analyses of the outcomes of interest will be masked from knowing the individuals' randomized treatment assignments, as will the principal investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group 1 (Active Comparator): Study Group 1 will begin the first treatment period with the provided Unfiltered Cigarettes intervention for two weeks, followed by a three-week wash-out period, before switching to the provided Filtered Cigarette intervention for two weeks.
  Interventions: Other: Unfiltered Cigarettes; Other: Filtered Cigarettes
- Study Group 2 (Experimental): Study Group 2 will begin the first treatment period with the provided Filtered Cigarettes intervention for two weeks, followed by a three-week wash-out period, before switching to the provided Unfiltered Cigarette intervention for two weeks.
  Interventions: Other: Unfiltered Cigarettes; Other: Filtered Cigarettes

INTERVENTIONS:
Other: Unfiltered Cigarettes — Participants will be given unfiltered Pall Mall or Camel cigarettes to smoke for two weeks according to the brand they smoked prior to the start of the study. They will agree to smoke the cigarettes using a monitoring device (CReSS) that measures puffing behavior on five (5) days during each of the two weeks. They will also collect their cigarette butts on all days as a measure of smoking behaviors.
Other: Filtered Cigarettes — Participants will be given filtered Pall Mall or Camel cigarettes to smoke for two weeks according to the brand they smoked prior to the start of the study. They will agree to smoke the cigarettes using a monitoring device (CReSS) that measures puffing behavior on five (5) days during each of the two weeks. They will also collect their cigarette butts on all days as a measure of smoking behaviors.

SUMMARY:
This study is an open-label, randomized, 9-week, two-sequence, two-treatment, cross-over clinical trial of 40 adult filtered cigarette smokers who switch to unfiltered cigarettes There will be a 1-week baseline period, 2 weeks of smoking filtered or unfiltered cigarettes (determined at time of randomization), and a 3-week washout period, followed by post-washout baseline week, and a crossover to 2 weeks of smoking the opposite condition.

DETAILED DESCRIPTION:
This innovative research project will assess the acceptability among committed smokers of switching to unfiltered cigarettes from filtered cigarettes and compare the measurement of exposure to nicotine and carcinogens after such a switch from filtered to unfiltered cigarettes. Such research will inform regulatory policy regarding the possibility of banning filters from the U.S. cigarette market. This high-impact pilot project is a randomized, cross-over clinical trial among smokers to measure changes in their puffing behavior, carcinogen exposures, nicotine exposure, and attitudes toward smoking unfiltered cigarettes if they were to no longer able to buy filtered cigarettes. The overall objective for this pilot trial is to collect preliminary data to inform design of a larger clinical trial in assessing changes in attitudes toward smoking unfiltered cigarettes; smoking topography; and urinary cotinine, urinary 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), and volatile organic compound (VOC) excretion resulting from switching from filtered to unfiltered cigarettes among a sample of committed smokers.

Aim 1. Determine smokers' satisfaction, and attitudes towards smoking cigarettes if they were to switch from smoking filtered to unfiltered cigarettes. The investigators hypothesize that smokers who smoke unfiltered cigarettes will have less satisfaction with their smoking compared with smoking filtered cigarettes.

Aim 2. Measure changes in smoking topography and cigarettes smoked per day among smokers who change to unfiltered cigarettes for two weeks compared with these measures while smoking filtered cigarettes. The investigators hypothesize that smokers who smoke unfiltered cigarettes for two weeks will change their topography such that they will inhale less deeply and frequently and will smoke fewer cigarettes per day.

Aim 3. Measure changes in urinary cotinine, NNAL, and VOC excretion among smokers who smoke unfiltered cigarettes for two weeks compared to smoking filtered cigarettes.

The investigators hypothesize that smokers who smoke unfiltered cigarettes for two weeks will have lower urinary cotinine, NNAL, and VOC excretion compared with filtered cigarettes.

The results from this trial can inform a larger clinical trial that can be submitted to the National Institutes of Health/Food and Drug Administration to develop evidence on the potentially positive impact of removing plastic filters from commercial cigarettes. It will allow us to develop sound scientific methods to assess the topography of smoking and excretion of cotinine, tobacco-specific nitrosamines, and VOCs by smokers who smoke cigarettes with and without filters. This new knowledge may lead the Food and Drug Administration or specific states to consider banning the sale of filtered cigarettes because filters make it easier for young people to start smoking, unjustifiably discourage smokers from quitting, and contaminate the environment with non-biodegradable, toxic waste.

ELIGIBILITY:
Inclusion Criteria:

* Are non-institutionalized, and
* Able to provide informed consent, and
* Are ages 21 to 65, and
* Smoke at least 25 days per month, and
* Smoke at least 5 cigarettes per day on the days they smoke, and
* Have been smoking cigarettes for at least 1 year, and
* Have smoked exclusively Camel or Pall Mall cigarettes over the past two weeks, or are willing to do so for the two weeks prior to, and for seven weeks during, the study, and
* Are fluent in English, and
* Have regular access to a telephone, and
* Have smoked only filtered cigarettes for the past year, and
* Have access to transportation to California State University, San Marcos (CSUSM), and
* Report primary (≥50% of the time) smoking of cigarettes, allowing for secondary use of other tobacco products, and
* Agree to the terms of the trial

Exclusion Criteria:

* Do not meet one or more of the above inclusion criteria, or
* Self-report uncontrolled diabetes (i.e., diagnosed with diabetes, and it is not being managed by a physician), or
* Present to the enrollment visit with a systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure greater than 105 mm Hg, or
* Self-report involvement in another clinical trial, or
* Self-report hospitalization for psychiatric issues or had a heart-related event (e.g. heart attack) at enrollment or within the past 30 days, or
* Self-report attempts to quit or cut down on smoking in past 30 days, or
* Self-report use of pharmacotherapy to aid smoking cessation within the past 30 days, or
* Are breastfeeding, pregnant, or may become pregnant during the next six months, or
* Are planning to move out of San Diego in the next 9 weeks, or
* Do not meet expected expired carbon monoxide (CO) measurements of smokers (Expired CO measurements>10 parts per million (ppm) will confirm status as a current smoker of at >5 cigarettes/day on the initial visit), or
* Are deemed mentally unstable (i.e., psychotic, under influence of drugs or alcohol, or unable to comprehend the call or meeting) or physically unfit (i.e, physically unwell) to participate in the study based on the researcher's determination at the enrollment visit

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mean flow rate (mL/s) | 9 weeks
  Mean flow rate, in mL per second, measures the flow of air through the CReSS as participants smoke cigarettes.
Change in number of puffs per cigarette | 9 weeks
  Measured by the CReSS device as participants smoke cigarettes
Change in duration of each cigarette puff (in seconds) | 9 weeks
  Measured by the CReSS device as participants smoke cigarettes
Change in inter-puff interval in seconds | 9 weeks
  The time between puffs on the cigarette, measured by the CReSS device as participants smoke cigarettes
Change in volume of each puff (mL) | 9 weeks
  Measured by the CReSS device as participants smoke cigarettes
Change in total smoke intake (mL) | 9 weeks
  Measured by the CReSS device as participants smoke cigarettes

SECONDARY OUTCOMES:
Urinary biomarker measurements | 9 weeks
  Target analytes are creatinine (the main proximate metabolite of nicotine), total (free + conjugated) 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (tNNAL, a carcinogenic tobacco-specific n-nitrosamine metabolite specific to tobacco smoke exposure), and a set of eight volatile organic compounds (VOCs, potentially toxic by-products of tobacco combustion). VOC concentrations will be measured at baseline in this study to account for possible additional sources of VOC exposure (assuming subjects' additional exposure remains consistent). VOCs will be measured as their urinary metabolites; i.e., mercapturic acid derivatives. The target parent VOCs are ethylene oxide, 1,3 butadiene, crotonaldehyde, acrolein, benzene, acrylamide, acrylonitrile, and propylene oxide. The biomarkers' urine concentration will be normalized to creatinine. Baseline midstream urine samples of at least 30 mL will be collected at baseline, post-washout, and at the end of each study cigarette period.
Cigarette satisfaction: mCEQ | 9 weeks
  Satisfaction with test cigarettes will be assessed using the 12-item modified Cigarette Evaluation Scale (mCEQ). This validated tool uses visual analog scales to assess subjective ratings: general acceptability ("bad" to "very good"), smoking need ("not at all" to "very strong"), smoking satisfaction ("not at all" to "very good"), harshness ("not at all" to "very strong") and pleasantness of smoke taste ("not tasty at all" to "very tasty"). Open-ended questions will also be asked regarding subject's experience smoking unfiltered cigarettes.
Change in answers to Stanford Perceptions Survey of Youth questions | 9 weeks
  Qualitative questions assessing knowledge abut cigarette filters, behaviors if filtered cigarettes were no longer available, and support for policy related to filtered cigarettes.
Change in perceptions of cigarette harshness | 9 weeks
  As measured by a visual analog scale of 0 (not harsh at all) to 100 (extremely harsh)
Change in perceptions of cigarette draw | 9 weeks
  As measured by a visual analog scale of 0 (very hard to draw smoke) to 100 (very easy to draw smoke)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Oren, Ph.D., Principal Investigator — San Diego State University School of Public Health; Kimberly Pulvers, Ph.D., Study Director — California State University, San Marcos
Locations (1):
- California State University San Marcos, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD), including a data dictionary, will be shared with the study's Data Safety and Monitoring Board (DSMB), or potentially with other collaborators in the future. It is not yet determined if there will be a plan to make the IPD available.

REFERENCES:
- [Background] Hastrup JL, Cummings KM, Swedrock T, Hyland A, Pauly JL. Consumers' knowledge and beliefs about the safety of cigarette filters. Tob Control. 2001 Mar;10(1):84. doi: 10.1136/tc.10.1.84. No abstract available. PMID 11347536
- [Background] Ito H, Matsuo K, Tanaka H, Koestler DC, Ombao H, Fulton J, Shibata A, Fujita M, Sugiyama H, Soda M, Sobue T, Mor V. Nonfilter and filter cigarette consumption and the incidence of lung cancer by histological type in Japan and the United States: analysis of 30-year data from population-based cancer registries. Int J Cancer. 2011 Apr 15;128(8):1918-28. doi: 10.1002/ijc.25531. PMID 20589676
- [Background] Brooks DR, Austin JH, Heelan RT, Ginsberg MS, Shin V, Olson SH, Muscat JE, Stellman SD. Influence of type of cigarette on peripheral versus central lung cancer. Cancer Epidemiol Biomarkers Prev. 2005 Mar;14(3):576-81. doi: 10.1158/1055-9965.EPI-04-0468. PMID 15767332
- [Background] Song MA, Benowitz NL, Berman M, Brasky TM, Cummings KM, Hatsukami DK, Marian C, O'Connor R, Rees VW, Woroszylo C, Shields PG. Cigarette Filter Ventilation and its Relationship to Increasing Rates of Lung Adenocarcinoma. J Natl Cancer Inst. 2017 Dec 1;109(12):djx075. doi: 10.1093/jnci/djx075. PMID 28525914
- [Background] Novotny TE, Slaughter E. Tobacco Product Waste: An Environmental Approach to Reduce Tobacco Consumption. Curr Environ Health Rep. 2014 May 6;1(3):208-216. doi: 10.1007/s40572-014-0016-x. eCollection 2014. PMID 25152862
- [Background] Slaughter E, Gersberg RM, Watanabe K, Rudolph J, Stransky C, Novotny TE. Toxicity of cigarette butts, and their chemical components, to marine and freshwater fish. Tob Control. 2011 May;20 Suppl 1(Suppl_1):i25-9. doi: 10.1136/tc.2010.040170. PMID 21504921
- [Background] Thun MJ, Carter BD, Feskanich D, Freedman ND, Prentice R, Lopez AD, Hartge P, Gapstur SM. 50-year trends in smoking-related mortality in the United States. N Engl J Med. 2013 Jan 24;368(4):351-64. doi: 10.1056/NEJMsa1211127. PMID 23343064
- [Background] Connolly GN, Alpert HR. Has the tobacco industry evaded the FDA's ban on 'Light' cigarette descriptors? Tob Control. 2014 Mar;23(2):140-5. doi: 10.1136/tobaccocontrol-2012-050746. Epub 2013 Mar 13. PMID 23485704
- [Background] Harris B. The intractable cigarette 'filter problem'. Tob Control. 2011 May;20 Suppl 1(Suppl_1):i10-6. doi: 10.1136/tc.2010.040113. PMID 21504917
- [Background] Czoli CD, Hammond D. Cigarette packaging: Youth perceptions of "natural" cigarettes, filter references, and contraband tobacco. J Adolesc Health. 2014 Jan;54(1):33-9. doi: 10.1016/j.jadohealth.2013.07.016. Epub 2013 Sep 4. PMID 24012064
- [Background] Samet JM, Aladadyan L. Should the FDA Ban Cigarette Filter Ventilation? J Natl Cancer Inst. 2017 Dec 1;109(12):djx073. doi: 10.1093/jnci/djx073. No abstract available. PMID 28525913
- [Background] Djordjevic MV, Stellman SD, Zang E. Doses of nicotine and lung carcinogens delivered to cigarette smokers. J Natl Cancer Inst. 2000 Jan 19;92(2):106-11. doi: 10.1093/jnci/92.2.106. PMID 10639511
- [Background] Pauly JL, Mepani AB, Lesses JD, Cummings KM, Streck RJ. Cigarettes with defective filters marketed for 40 years: what Philip Morris never told smokers. Tob Control. 2002 Mar;11 Suppl 1(Suppl 1):I51-61. doi: 10.1136/tc.11.suppl_1.i51. PMID 11893815
- [Background] Novotny TE, Hardin SN, Hovda LR, Novotny DJ, McLean MK, Khan S. Tobacco and cigarette butt consumption in humans and animals. Tob Control. 2011 May;20 Suppl 1(Suppl_1):i17-20. doi: 10.1136/tc.2011.043489. PMID 21504918
- [Background] Oren E, Bell ML, Garcia F, Perez-Velez C, Gerald LB. Promoting adherence to treatment for latent TB infection through mobile phone text messaging: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2017 Mar 13;3:15. doi: 10.1186/s40814-017-0128-9. eCollection 2017. PMID 28293431
- [Background] Horne DJ, Campo M, Ortiz JR, Oren E, Arentz M, Crothers K, Narita M. Association between smoking and latent tuberculosis in the U.S. population: an analysis of the National Health and Nutrition Examination Survey. PLoS One. 2012;7(11):e49050. doi: 10.1371/journal.pone.0049050. Epub 2012 Nov 8. PMID 23145066
- [Background] Oren E, Rothers J, Stern DA, Morgan WJ, Halonen M, Wright AL. Cough during infancy and subsequent childhood asthma. Clin Exp Allergy. 2015 Sep;45(9):1439-46. doi: 10.1111/cea.12573. PMID 26011047
- [Background] Matt GE, Quintana PJE, Zakarian JM, Hoh E, Hovell MF, Mahabee-Gittens M, Watanabe K, Datuin K, Vue C, Chatfield DA. When smokers quit: exposure to nicotine and carcinogens persists from thirdhand smoke pollution. Tob Control. 2016 Sep;26(5):548-556. doi: 10.1136/tobaccocontrol-2016-053119. Epub 2016 Sep 21. PMID 27655249
- [Background] Matt GE, Quintana PJE, Hoh E, Zakarian JM, Chowdhury Z, Hovell MF, Jacob P, Watanabe K, Theweny TS, Flores V, Nguyen A, Dhaliwal N, Hayward G. A Casino goes smoke free: a longitudinal study of secondhand and thirdhand smoke pollution and exposure. Tob Control. 2018 Nov;27(6):643-649. doi: 10.1136/tobaccocontrol-2017-054052. Epub 2018 Feb 8. PMID 29439207
- [Background] Matt GE, Quintana PJ, Fortmann AL, Zakarian JM, Galaviz VE, Chatfield DA, Hoh E, Hovell MF, Winston C. Thirdhand smoke and exposure in California hotels: non-smoking rooms fail to protect non-smoking hotel guests from tobacco smoke exposure. Tob Control. 2014 May;23(3):264-72. doi: 10.1136/tobaccocontrol-2012-050824. Epub 2013 May 13. PMID 23669058
- [Background] Pulvers K, Hood A, Limas EF, Thomas MD. Female smokers show lower pain tolerance in a physical distress task. Addict Behav. 2012 Oct;37(10):1167-70. doi: 10.1016/j.addbeh.2012.05.002. Epub 2012 May 22. PMID 22658302
- [Background] Pulvers K, Emami AS, Nollen NL, Romero DR, Strong DR, Benowitz NL, Ahluwalia JS. Tobacco Consumption and Toxicant Exposure of Cigarette Smokers Using Electronic Cigarettes. Nicotine Tob Res. 2018 Jan 5;20(2):206-214. doi: 10.1093/ntr/ntw333. PMID 28003511
- [Background] Morabia A, Bernstein MS, Curtin F, Berode M. Validation of self-reported smoking status by simultaneous measurement of carbon monoxide and salivary thiocyanate. Prev Med. 2001 Jan;32(1):82-8. doi: 10.1006/pmed.2000.0779. PMID 11162330
- [Background] Ripoll J, Girauta H, Ramos M, Medina-Bombardo D, Pastor A, Alvarez-Ossorio C, Gorreto L, Esteva M, Garcia E, Urendez A, Buades A, Torres E. Clinical trial on the efficacy of exhaled carbon monoxide measurement in smoking cessation in primary health care. BMC Public Health. 2012 Jul 4;12:322. doi: 10.1186/1471-2458-12-322. PMID 22551017
- [Background] Javors MA, Hatch JP, Lamb RJ. Cut-off levels for breath carbon monoxide as a marker for cigarette smoking. Addiction. 2005 Feb;100(2):159-67. doi: 10.1111/j.1360-0443.2004.00957.x. PMID 15679745
- [Background] Zhu SH, Pulvers K, Zhuang Y, Baezconde-Garbanati L. Most Latino smokers in California are low-frequency smokers. Addiction. 2007 Oct;102 Suppl 2:104-11. doi: 10.1111/j.1360-0443.2007.01961.x. PMID 17850620
- [Background] Rahmanian SD, Diaz PT, Wewers ME. Tobacco use and cessation among women: research and treatment-related issues. J Womens Health (Larchmt). 2011 Mar;20(3):349-57. doi: 10.1089/jwh.2010.2173. PMID 21375414
- [Background] Cubbin C, Soobader MJ, LeClere FB. The intersection of gender and race/ethnicity in smoking behaviors among menthol and non-menthol smokers in the United States. Addiction. 2010 Dec;105 Suppl 1:32-8. doi: 10.1111/j.1360-0443.2010.03191.x. PMID 21059134
- [Background] Weinberger AH, McKee SA. Mood and smoking behavior: the role of expectancy accessibility and gender. Addict Behav. 2012 Dec;37(12):1349-52. doi: 10.1016/j.addbeh.2012.07.010. Epub 2012 Jul 28. PMID 22958868
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Hammond D, Fong GT, Cummings KM, O'Connor RJ, Giovino GA, McNeill A. Cigarette yields and human exposure: a comparison of alternative testing regimens. Cancer Epidemiol Biomarkers Prev. 2006 Aug;15(8):1495-501. doi: 10.1158/1055-9965.EPI-06-0047. PMID 16896039
- [Background] Blank MD, Disharoon S, Eissenberg T. Comparison of methods for measurement of smoking behavior: mouthpiece-based computerized devices versus direct observation. Nicotine Tob Res. 2009 Jul;11(7):896-903. doi: 10.1093/ntr/ntp083. Epub 2009 Jun 11. PMID 19525207
- [Background] Gust SW, Pickens RW. Does cigarette nicotine yield affect puff volume? Clin Pharmacol Ther. 1982 Oct;32(4):418-22. doi: 10.1038/clpt.1982.182. No abstract available. PMID 7116755
- [Background] Zacny JP, Stitzer ML. Effects of smoke deprivation interval on puff topography. Clin Pharmacol Ther. 1985 Jul;38(1):109-15. doi: 10.1038/clpt.1985.143. PMID 4006371
- [Background] Lee EM, Malson JL, Waters AJ, Moolchan ET, Pickworth WB. Smoking topography: reliability and validity in dependent smokers. Nicotine Tob Res. 2003 Oct;5(5):673-9. doi: 10.1080/1462220031000158645. PMID 14577984
- [Background] Blank MD, Breland AB, Enlow PT, Duncan C, Metzger A, Cobb CO. Measurement of smoking behavior: Comparison of self-reports, returned cigarette butts, and toxicant levels. Exp Clin Psychopharmacol. 2016 Oct;24(5):348-355. doi: 10.1037/pha0000083. Epub 2016 Jun 27. PMID 27347741
- [Background] Clark PI, Gautam SP, Hlaing WM, Gerson LW. Response error in self-reported current smoking frequency by black and white established smokers. Ann Epidemiol. 1996 Nov;6(6):483-9. doi: 10.1016/s1047-2797(96)00049-x. PMID 8978878
- [Background] Wye P, Gow LB, Constable J, Bowman J, Lawn S, Wiggers J. Observation of the extent of smoking in a mental health inpatient facility with a smoke-free policy. BMC Psychiatry. 2014 Mar 29;14:94. doi: 10.1186/1471-244X-14-94. PMID 24679109
- [Background] Goniewicz ML, Havel CM, Peng MW, Jacob P 3rd, Dempsey D, Yu L, Zielinska-Danch W, Koszowski B, Czogala J, Sobczak A, Benowitz NL. Elimination kinetics of the tobacco-specific biomarker and lung carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol. Cancer Epidemiol Biomarkers Prev. 2009 Dec;18(12):3421-5. doi: 10.1158/1055-9965.EPI-09-0874. PMID 19959691
- [Background] Jacob P 3rd, Havel C, Lee DH, Yu L, Eisner MD, Benowitz NL. Subpicogram per milliliter determination of the tobacco-specific carcinogen metabolite 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol in human urine using liquid chromatography-tandem mass spectrometry. Anal Chem. 2008 Nov 1;80(21):8115-21. doi: 10.1021/ac8009005. Epub 2008 Oct 8. PMID 18841944
- [Background] Jain RB. Levels of selected urinary metabolites of volatile organic compounds among children aged 6-11 years. Environ Res. 2015 Oct;142:461-70. doi: 10.1016/j.envres.2015.07.023. Epub 2015 Aug 7. PMID 26257031
- [Background] Goniewicz ML, Gawron M, Smith DM, Peng M, Jacob P 3rd, Benowitz NL. Exposure to Nicotine and Selected Toxicants in Cigarette Smokers Who Switched to Electronic Cigarettes: A Longitudinal Within-Subjects Observational Study. Nicotine Tob Res. 2017 Feb;19(2):160-167. doi: 10.1093/ntr/ntw160. Epub 2016 Aug 17. PMID 27613896
- [Background] Dodder NG, Tai SS, Sniegoski LT, Zhang NF, Welch MJ. Certification of creatinine in a human serum reference material by GC-MS and LC-MS. Clin Chem. 2007 Sep;53(9):1694-9. doi: 10.1373/clinchem.2007.090027. Epub 2007 Jul 27. PMID 17660272
- [Background] Tonstad S, Gustavsson G, Kruse E, Walmsley JM, Westin A. Symptoms of nicotine toxicity in subjects achieving high cotinine levels during nicotine replacement therapy. Nicotine Tob Res. 2014 Sep;16(9):1266-71. doi: 10.1093/ntr/ntu076. Epub 2014 May 22. PMID 24852574
- [Background] Jacob P 3rd, Yu L, Duan M, Ramos L, Yturralde O, Benowitz NL. Determination of the nicotine metabolites cotinine and trans-3'-hydroxycotinine in biologic fluids of smokers and non-smokers using liquid chromatography-tandem mass spectrometry: biomarkers for tobacco smoke exposure and for phenotyping cytochrome P450 2A6 activity. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Feb 1;879(3-4):267-76. doi: 10.1016/j.jchromb.2010.12.012. Epub 2010 Dec 21. PMID 21208832
- [Background] Benowitz NL, Dains KM, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Progressive commercial cigarette yield reduction: biochemical exposure and behavioral assessment. Cancer Epidemiol Biomarkers Prev. 2009 Mar;18(3):876-83. doi: 10.1158/1055-9965.EPI-08-0731. Epub 2009 Mar 3. PMID 19258480
- [Background] Benowitz NL, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Nicotine and carcinogen exposure with smoking of progressively reduced nicotine content cigarette. Cancer Epidemiol Biomarkers Prev. 2007 Nov;16(11):2479-85. doi: 10.1158/1055-9965.EPI-07-0393. PMID 18006940
- [Derived] Pulvers K, Tracy L, Novotny TE, Satybaldiyeva N, Hunn A, Romero DR, Dodder NG, Magraner J, Oren E. Switching people who smoke to unfiltered cigarettes: perceptions, addiction and behavioural effects in a cross-over randomised controlled trial. Tob Control. 2023 Jul;32(4):520-523. doi: 10.1136/tobaccocontrol-2021-056815. Epub 2021 Nov 19. PMID 34799433
- [Derived] Oren E, Pulvers K, Romero DR, Barber C, Carter E, Tracy LA, Novotny TE. Effects of Unfiltered Cigarettes on Smoking Behavior and Toxicant Exposure: Protocol for a Randomized Crossover Clinical Trial. JMIR Res Protoc. 2020 Dec 8;9(12):e19603. doi: 10.2196/19603. PMID 33289680